CLINICAL TRIAL: NCT05455710
Title: Evaluation of Post-discharge Surveillance Mobile Application for Surgical Site Infection as a Clinical Decision Support System
Brief Title: Evaluation of Post-discharge Surveillance Mobile Application for Surgical Site Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Camila Dalcól, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Vigi-App
Record Dates: First submitted 2020-10-09; First posted 2022-07-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Surgical Wound Infection
Keywords: Mobile applications; Patient discharge; Surgical wound infection; Public health surveillance; Perioperative nursing.
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: In order to verify the effectiveness of the mobile application for post-discharge surveillance the developed infection of the surgical site, a randomized clinical trial of superiority will be carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VigiApp (Experimental): the intervention group, which will use the mobile application to detect SSI. The Vigi-App application will be installed on the Smartphone of the selected patients, who will receive training on how to use the application; should access it on days seven, 14, 21 and 30 after the surgical procedure, they will additionally be evaluated in person in an outpatient consultation, according to the hospital routine.
  The patients in the intervention group will receive notices the day before, through reminders issued by the application, reminding them that they must access and complete the requested information. If the patient presents signs and symptoms of infection on dates other than filling out the application, he can access the application and send his data normally as an extra access.
  Interventions: Device: VigiApp
- telephone call (Sham Comparator): the called control, consisting of the standard infection surgical site post-discharge surveillance the developed infection of the surgical site procedure, by means of a telephone call. You will receive guidance on phone calls; will follow the standard SSI post-discharge surveillance procedure, by means of a telephone call on days seven, 14, 21 and 30 after the date of surgery, being asked about the presence of signs and symptoms of infection according to the instrument previously validated in previous investigation and will be evaluated in person in an outpatient consultation, according to the hospital routine.
  Interventions: Device: VigiApp

INTERVENTIONS:
Device: VigiApp — mobile application containing a patient identification module; post-discharge surveillance questionnaire with questions related to signs and symptoms of SSI previously validated; possibility of attaching and sending a photograph of the surgical wound; field for exchanging messages between professional and patient; issuing an alert / reminder to fill in the data in the application; in addition to establishing interoperability with the system used by the hospital's SCIH, containing a login for each health professional, which allows access to the answers, images and messages sent by surgical patients, categorizing risk and issuing alerts in suspected cases of SSI.

SUMMARY:
Objective: evaluate the effectiveness and usability of a mobile application for post-discharge surveillance of surgical site infection as a support system for clinical decision.

DETAILED DESCRIPTION:
Introduction: Infection of the surgical site (SSI) is one of the main infections related to health care, culminating in financial losses to the health system and high morbidity and mortality, which due to increasingly shorter hospital stays, from 13 to 75% is manifested at home of the patient, requiring health professionals to act more effectively in post-discharge surveillance of this condition. Therefore, considering this problem and the constant evolution of technological resources, with the increase in access and use of smartphones by the population, it is pertinent to develop a mobile application for post-discharge surveillance of surgical site infection. Objective: evaluate the effectiveness and usability of a mobile application for post-discharge surveillance of surgical site infection as a support system for clinical decision. Method: Randomized Clinical Trial to assess effectiveness of a mobile application for post-discharge surveillance of infection of the surgical site. The study will be developed in a large hospital in the city of São Paulo and the study participants will be surgical patients. Expected results: The mobile application for post-discharge surveillance is expected to collaborate in the early detection of potential cases of surgical site infection, to be able to improve post-discharge surveillance strategies, assist in data management, decision making and actions to prevent infection of the surgical site.

ELIGIBILITY:
Inclusion Criteria:

* surgical patients aged 18 to 70 years
* conscious, oriented,
* literate
* have a smartphone compatible with the use of the application
* submitted to traditional anesthetic-surgical procedure
* classified as potentially contaminated
* experience the postoperative period at home

Exclusion Criteria:

* Patients with visual impairment
* physical restriction or communication problems
* undergoing surgery with implants
* videolaparoscopies or robotics sugery
* who already have the diagnosis of SSI at the time of discharge
* have been admitted to the Intensive Care Unit in the postoperative period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
effectiveness of the mobile app - sensitivity | Four months
  The effectiveness of the integrated mobile application for the SSI post-discharge surveillance in the correct and early identification of the SSI, through measures of sensitivity in percentage.
effectiveness of the mobile app - specificity | Four months
  The effectiveness of the integrated mobile application for the SSI post-discharge surveillance in the correct and early identification of the SSI, through measures of specificity in percentage.

SECONDARY OUTCOMES:
rate of adherence | Four months
  The rate of adherence will be verified, quantitatively, according to the number of patients accessing the application and according to the successful telephone contact of healthcare professionals with patients.
usability and user satisfaction | Four months
  To assess usability and user satisfaction, the Measurement Inventory Usability Software will be used, in likert (agree and disagree), which 50 items, with user satisfaction in use in five usability dimensions: efficiency, satisfaction, usefulness , control and learning, each with 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Poveda, doutorate, Study Director — USP
Locations (2):
- Brazil (2):
  - Hospital Universitário UFSC, Florianópolis
  - ICESP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiseman JT, Fernandes-Taylor S, Barnes ML, Tomsejova A, Saunders RS, Kent KC. Conceptualizing smartphone use in outpatient wound assessment: patients' and caregivers' willingness to use technology. J Surg Res. 2015 Sep;198(1):245-51. doi: 10.1016/j.jss.2015.05.011. Epub 2015 May 14. PMID 26025626
- [Background] Sanger PC, Hartzler A, Han SM, Armstrong CA, Stewart MR, Lordon RJ, Lober WB, Evans HL. Patient perspectives on post-discharge surgical site infections: towards a patient-centered mobile health solution. PLoS One. 2014 Dec 1;9(12):e114016. doi: 10.1371/journal.pone.0114016. eCollection 2014. PMID 25436912
- [Background] Gunter RL, Fernandes-Taylor S, Rahman S, Awoyinka L, Bennett KM, Weber SM, Greenberg CC, Kent KC. Feasibility of an Image-Based Mobile Health Protocol for Postoperative Wound Monitoring. J Am Coll Surg. 2018 Mar;226(3):277-286. doi: 10.1016/j.jamcollsurg.2017.12.013. Epub 2018 Jan 19. PMID 29366555
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957